CLINICAL TRIAL: NCT05596461
Title: Research on New Techniques for Diagnosis and Treatment of Neuropsychiatric Diseases - Research on New Techniques for Diagnosis and Treatment of Affective Disorders and Cognitive Impairment
Brief Title: New Techniques for Diagnosis and Treatment of Cognitive Impairment in Affective Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, Head of Department of Psychaitry , First Affiliated Hospital of Zhejiang University, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT20210036C-R1
Record Dates: First submitted 2022-05-26; First posted 2022-10-27 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Affective Disorder
MeSH Terms: conditions — Mood Disorders | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial magnetic stimulation (Experimental)
  Interventions: Device: Transcranial magnetic stimulation
- Transcranial direct-current stimulation (Experimental)
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Setting up a new target for rTMS. In the past research, the common target of rTMS in the treatment of cognitive impairment of affective disorder was left Dorsolateral prefrontal CORTEX (DLPFC) . The left lateral DLPFC and the primary visual Cortex (V1) both play important roles in cognitive process. The regions with the strongest functional connection between V1 and DLPFC were selected as the stimulation targets.
  Arms: Transcranial magnetic stimulation
Device: Transcranial direct current stimulation — Targeted multi-channel tDCS based on individualized simulation scale can be combined with individualized simulation modeling optimization, and based on individual MRI information, through quantitative evaluation and intelligent algorithms to achieve stimulation parameter optimization, reduce the stimulation dose to non-target target areas, and improve target brain stimulation The treatment targeting and aggregation of the area can realize personalized and precise treatment.
  Arms: Transcranial direct-current stimulation

SUMMARY:
The purpose of this study is to explore the pathological mechanism of cognitive impairment in patients with affective disorder based on brain gut axis research, preliminarily verify the clinical efficacy of new neural regulation technology on cognitive impairment, and establish an evaluation model to predict the efficacy of physical therapy for affective disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-65 years old, regardless of gender;
2. Meet DSM-V diagnostic criteria for depression or bipolar disorder;
3. Duration of stable period ≥ 3 months;
4. Young Mania Rating Scale (YMRS) ≤ 6 points;
5. Hamilton Depression Rating Scale 17 - item (HDRS-17) score ≤ 7;
6. The score of cognitive defects questionnaire (PDQ) ≥ 17;
7. Han nationality, right-handed;
8. More than 9 years of education.

Exclusion Criteria:

1. History of severe somatic or brain organic diseases and craniocerebral trauma;
2. Abnormal brain structure or any MRI contraindications were found by magnetic resonance examination;
3. Those who do not cooperate or cannot effectively complete the experiment;
4. Drug, alcohol or other psychoactive substance abusers;
5. Pregnant, lactating or planned pregnancy.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Wechsler Memory Scale | 0-8 weeks
  The Wechsler Memory Scale score was used to evaluate the degree of cognitive function, and the lower the score, the more severe the cognitive function impairment. The scoring threshold is 70 points. A lower score means more severe cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhou H, Wang M, Xu T, Zhang X, Zhao X, Tang L, Zhao P, Wang D, Lai J, Wang F, Zhang S, Hu S. Cognitive Remediation in Patients With Bipolar Disorder: A Randomized Trial by Sequential tDCS and Navigated rTMS Targeting the Primary Visual Cortex. CNS Neurosci Ther. 2024 Dec;30(12):e70179. doi: 10.1111/cns.70179. PMID 39703101